CLINICAL TRIAL: NCT07282691
Title: Validation of Clinical Outcome Measures Specific to mTBI-Related Oculomotor Disorders
Status: Recruiting | Type: Observational
Sponsor: Salus University (Other)
Responsible Party: Sponsor
Other Study IDs: 2406010608
Record Dates: First submitted 2025-11-12; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: MTBI - Mild Traumatic Brain Injury
Keywords: mTBI; convergence insufficiency; concussion; concussion-related vision disorders; vision rehabilitation; vision therapy
MeSH Terms: conditions — Brain Concussion; Ocular Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control participants: no history of mTBI
- mTBI group: history of mTBI

SUMMARY:
The specific aim of this project is to validate clinical tests to be used as outcome measures in studies of mTBI-related vision problems.

DETAILED DESCRIPTION:
Participants with (n=50) and without (n=100) a history of mTBI will be recruited. Investigators will study the use of a series of visual endurance tests (tests that require sustained visual responses over a period of time). In addition to developing expected values for these tests, investigators will also after qualitative data about discomfort levels during testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mTBI within previous 1 to 6 months
* Distance visual acuity better than or equal to 20/25 in each eye
* Score >21 on Convergence Insufficiency Symptom Survey

Exclusion Criteria:

* Diagnosis of moderate or severe TBI; > 30-min loss of consciousness
* Not wearing required refractive error)
* Disease(s) known to affect oculomotor system (multiple sclerosis, Graves orbitopathy, myasthenia gravis, diabetes mellitus, or Parkinson disease)-Manifest strabismus or intraocular injury (evaluated at vision examination)
* Cognitive delays that may impact testing

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: mTBI
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-09-29 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with abnormal near point of convergence | Baseline and visit 2, which occurs 8 weeks after the baseline visit
  The ability to converge the eyes. A near point rod will be used with a 20/30 column of letters. The target will be moved towards the participant slowly, and when diplopia occurs, this will be recorded as the NPC break. The target will then be moved away from the eyes until single vision is regained, and this will be recorded as the NPC recovery. The unit of measure is cm and the NPC will be measured 3 times, with 10 seconds in between each measure, and averaged for each participant.

SECONDARY OUTCOMES:
Number of participants with abnormal positive fusional vergence | Baseline and visit 2, which occurs 8 weeks after the baseline visit
  Compensatory ability to overcome exophoria. A handheld prism bar will be used along with a vertical column of 20/30 letters. The prism will be placed before one eye, and the participant will be asked to maintain clear, single vision. Participants will then report when the target becomes blurred (blur), then double (diplopia), and finally return to single vision (recovery). The unit of measure is prism diopters, and it will be measured three times, with 10 seconds in between each measurement, and averaged for each participant.
Number of participants with abnormal vergence facility | Baseline and visit 2, which occurs 8 weeks after the baseline visit
  This is a measure of vergence velocity. Using a 12-base-out and 3-base-in prism, participants will be instructed to regain clear single vision as quickly as possible. The investigator will count the number of times this can be accomplished in one minut.e
Number of participants with abnormal accommodative amplitude | Baseline and visit 2, which occurs 8 weeks after the baseline visit
  A near point rod will be used along with a column of 20/30 letters. The test will be performed monocularly, first with the left eye covered, and then with the right eye covered. The target will slowly be moved towards the participant, and the participant will be instructed to report when the target becomes blurred. The amplitude of accommodation will be measured 3 times, with 10 seconds in between each measure
Number of participants with abnormal accommodative facility | Baseline and visit 2, which occurs 8 weeks after the baseline visit
  This test assesses the speed and endurance of accommodation. A column of 20/30 letter will be used along with a timer, and +2.00D and -2.00D lens flippers. The test will be performed monocularly. The +2.00D lens will be placed before the participant's eye, and the participant will be asked to clear the target as quickly as possible. Once the participant clears the target, the -2.00D lens will be placed before the eye, and the participant will be asked to report when the target becomes clear again. This will be repeated as many times as possible within one minute. The investigator will report how many times this occurs in one minute.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Scheiman, Study Chair — Pennsylvania College of Optometry at Drexel University
Locations (1):
- The Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The IPD will only be shared with the study investigators. REDCap will be used for data collection.